CLINICAL TRIAL: NCT06027060
Title: Observational Study on Monitoring NSAID-Induced Gastropathy in Patients Using Magnetically-Controlled Capsule Gastroscopy
Status: Suspended | Type: Observational
Why Stopped: Failure of equipment
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Renjixh202301
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: NSAID-Associated Gastropathy
Keywords: Magnetically-controlled Capsule Endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSAIDs users: 90 patients taking NSAIDs for over 3 months
- non-NSAIDs users: 90 non-NSAIDs users undergoing physical examination

SUMMARY:
The objective of this study is to observe gastric mucosal injuries in NSAID and non-NSAID users with magnetically-controlled capsule gastroscopy, and explore the effects of NSAIDs on gastric mucosal damage.

DETAILED DESCRIPTION:
Non-steroidal anti-inflammatory drugs are widely used in all kinds of people in China. A major limitation to their use is the adverse effects they cause on the gastrointestinal tract, including the formation of stomach lesions, ulcers due to stress reactions, and damage to the healing of gastric ulcers. The purpose of this prospective, single-center study was to monitor the gastric mucosal injury in patients with and without NSAIDs using magnetron capsule gastroscopy, and to explore the effect of NSaids on gastric mucosal injury.

For people taking NSAIDs, it is necessary to regularly detect gastric mucosal damage, and timely intervention treatment is required if relevant lesions are found, and the medication plan is adjusted. Magnetron capsule gastroscope has the advantages of comfort, safety, no anesthesia, no risk of cross infection, etc. It is highly accepted by the population, and is a beneficial supplement to traditional gastroscopy, so that some people with absolute or relative contraindications of traditional gastroscopy can get timely endoscopy, and can be diagnosed and treated early.

ELIGIBILITY:
Inclusion Criteria:

* Planned magnetically-controlled capsule gastroscopy
* NSAID use >3 months or no NSAID use
* Informed consent

Exclusion Criteria:

* No surgical conditions or refuses abdominal surgery (Once the capsule is stuck it cannot be removed surgically);
* Cardiac pacemakers (except MRI-compatible ones);
* Electronic implants or metal foreign bodies;
* Pregnant women;
* Known or suspected GI obstruction, stenosis, fistula;
* Dysphagia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ninety patients receiving NSAIDS (more than 3 months) and undergoing magnetron capsule gastroscopy at Renji Hospital were included, and 90 patients not taking NSAIDS and undergoing magnetron capsule gastroscopy at the same time were included.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Gastric diseases detected | 1 day
  Gastric diseases detected

SECONDARY OUTCOMES:
Gastric mucosal injury by Lanza score | 1 day
  Gastric mucosal injury by Lanza score
Gastric transit time | 1 day
  Gastric transit time
Gastric cleanliness | 1 day
  Gastric cleanliness
Effects of NSAID duration on gastric injury | 1 day
  Effects of NSAID duration on gastric injury
Effects of NSAID dosage on gastric injury | 1 day
  Effects of NSAID dosage on gastric injury

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No